CLINICAL TRIAL: NCT01152320
Title: Randomized Controlled Trial of Spirometry Fundamentals™ in the Primary Care Setting
Brief Title: Trial of Spirometry Fundamentals™ in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Rita Mangione-Smith, University of Washington/Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 31552-E/A; A26829 (Other Grant/Funding Number: American Thoracic Society)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Asthma
Keywords: Asthma; Spirometry; Pediatric; Primary Health Care; Education, Distance
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention)
- Intervention (Experimental): Spirometry Fundamentals™ CD training program
  Interventions: Behavioral: Spirometry Fundamentals™ Training CD

INTERVENTIONS:
Behavioral: Spirometry Fundamentals™ Training CD — MD-MA pairs randomized to the intervention arm of the study received 2 copies of the Spirometry Fundamentals™ CD. Included with the CDs was a letter explaining that each member of the MD-MA pair should view the CD at their convenience within the following 3 weeks. This letter included instructions on how to access the study website in order to complete an evaluation survey after viewing the CD.
  Arms: Intervention

SUMMARY:
Spirometry is a recommended component of asthma diagnosis and treatment in the primary care setting, yet few primary care providers report routine use of spirometry in the provision of care for their asthma patients. Misclassification of asthma severity has been reported when assessment is based on symptoms alone. This misclassification can lead to inadequate treatment that may result in increased morbidity and increased healthcare utilization/cost. However, even when spirometry is utilized to aid in asthma severity classification, primary care providers have a high rate of failing to meet the quality goals for testing established by the American Thoracic Society.

The goal of this study is to evaluate the effectiveness of the Spirometry Fundamentals™ tool in training primary care providers and their staff in producing high-quality flow-volume curves as compared to existing training modalities and to gather information in a 'real-world' setting that can be used to improve Spirometry Fundamentals™.

DETAILED DESCRIPTION:
Currently few self-paced, distance learning programs exist that train staff to perform good quality spirometry tests. This study evaluates the effectiveness of a distance-learning tool for training primary care providers and their medical assistants in the use of spirometry to assist in managing obstructive lung disease (asthma and COPD). This tool is called "Spirometry Fundamentals™: A basic guide to lung function testing". It is a computer-based training program that teaches primary care providers and their staff what spirometry is, how it can be used, the techniques required to perform high-quality spirometry, and clinical interpretation of the spirometric data.

We evaluated the effectiveness of Spirometry Fundamentals in the primary care setting by conducting a randomized controlled trial (RCT). Study participants were primary care physicians (MDs or DOs) and their staff (medical assistants (MAs) or nurses (RNs)) and were recruited as study pairs. The role of the MDs was to utilize spirometry in clinical care by ordering spirometry tests based on their clinical judgment, and the role of the MAs was to perform the spirometry. The patients performed the spirometry as part of their usual care were not considered study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have internet access in order to transmit spirometry curve and survey data.
* Subjects must have access to a computer with Windows 2000 /Mac OS 10 or higher in order to view Spirometry Fundamentals™.
* Subjects must have access to a ndd Easyone spirometer.

Exclusion Criteria:

* Subjects who lack internet access which will be needed to transmit study data
* Subjects who lack access to a computer with Windows 2000 /Mac OS 10 or higher which will be needed to view Spirometry Fundamentals™.
* Subjects who lack access to a ndd Easyone spirometer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Spirometry test quality | Four months for controls; six months for intervention sites
  Percentage of acceptable quality spirometry tests as determined by standards set by the American Thoracic Society.

SECONDARY OUTCOMES:
Effect of frequency of spirometry use on primary outcome | Four months for controls; six months for intervention sites
  Examined whether frequency of spirometry use related to the percent of passing testing sessions conducted by the office.
Effect of practice location on primary outcome | Four months for controls; six months for intervention sites
  Examined whether practice location (private/community, hospital/university) related to the percent of passing testing sessions conducted by the office.
Effect of practice type on primary outcome | Four months for controls; six months for intervention sites
  Examined whether practice type (pediatric/non-pediatric) related to the percent of passing testing sessions conducted by the office.
Effect of practice structure on primary outcome | Four months for controls; six months for intervention sites
  Examined whether practice structure related to the percent of passing testing sessions conducted by the office.
Effect of months of spirometry use on primary outcome | Four months for controls; six months for intervention sites
  Examined whether months of spirometry use by practice (prior to participating in study) related to the percent of passing testing sessions conducted by the office.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mangione-Smith, MD, MPH, Principal Investigator — University of Washington/Seattle Children's Hospital; James W Stout, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: Site for primary care physicians to learn about Spirometry — http://www.spirometrytraining.org/